CLINICAL TRIAL: NCT07263399
Title: Effect of Hydrogen Gas on Hyperbaric Oxygen Toxicity - A Randomized Controlled Cross-Over Trial
Brief Title: Effect of Hydrogen Gas on Hyperbaric Oxygen Toxicity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blekinge Institute of Technology (Other)
Collaborators: Karolinska Institutet (Other); Göteborg University (Other); Lund University (Other); Swedish Armed Forces Diving and Naval Medicine Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BTH-6.1.1-0165-2025; 5005113/22FMV2951 (Other Grant/Funding Number: Swedish Armed Forces Material Administration)
Record Dates: First submitted 2025-09-29; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Oxygen Toxicity; Oxidative Stress; Hyperoxia; Hyperbaric Oxygen; Healthy Subjects (HS); Diving Medicine; Hydrogen-oxygen Gas
Keywords: Pulmonary Oxygen Toxicity; Hydrogen Gas; Diving Physiology; Lung Function; Hyperbaric Oxygen; Human Study; Military Divers
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Intervention Model Description: This is a human randomized, double-blind, crossover trial in which each participant undergoes two separate hyperbaric oxygen exposures: one with hydrogen-enriched breathing gas (1-2% H₂) and one with nitrogen-enriched breathing gas (1-2% N₂) as control. Before and after each exposure session, participants complete standardized pulmonary function tests and provide blood and urin samples for analysis of oxidative stress biomarkers. A washout period of at least two weeks is maintained between sessions to minimize carryover effects.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen Gas Intervention (Experimental): In this arm, participants will undergo a single hyperbaric exposure breathing a gas mixture composed of 98-99% oxygen and 1-2% hydrogen (H₂) at a partial pressure of 1.75 ATA for 240 minutes. The intervention aims to evaluate whether hydrogen gas has protective effects against pulmonary oxygen toxicity. Pulmonary function tests and blood and urin sampling for oxidative stress biomarkers will be performed both before and after the exposure session. The order of intervention and control exposures is randomized and the study is conducted in a double-blind fashion.
  A washout period of at least two weeks will follow before the control
  Interventions: Other: Inhaled Hydrogen-Enriched Oxygen Gas; Other: Inhaled Nitrogen-Enriched Oxygen Gas
- Nitrogen Gas Control (Active Comparator): In this arm, participants will undergo a single hyperbaric exposure breathing a gas mixture composed of 98-99% oxygen and 1-2% nitrogen (N₂) at a partial pressure of 1.75 ATA for 240 minutes. This exposure serves as the control condition and represents the standard oxygen-enriched breathing gas currently in use. Pulmonary function tests and blood and urin sampling for oxidative stress biomarkers will be performed both before and after the exposure session. Participants will be randomized to the order of exposures, and both participants and investigators will be blinded to the gas composition. A washout period of at least two weeks will follow before the intervention.
  Interventions: Other: Inhaled Hydrogen-Enriched Oxygen Gas; Other: Inhaled Nitrogen-Enriched Oxygen Gas

INTERVENTIONS:
Other: Inhaled Hydrogen-Enriched Oxygen Gas — Participants will inhale a gas mixture consisting of 98-99% oxygen and 1-2% hydrogen via a breathing circuit during a single hyperbaric exposure. The exposure will be conducted at a partial pressure of 1.75 ATA for 240 minutes. The intervention aims to evaluate the protective effect of hydrogen gas against pulmonary oxygen toxicity.
Other: Inhaled Nitrogen-Enriched Oxygen Gas — Participants will inhale a gas mixture consisting of 98-99% oxygen and 1-2% nitrogen via a breathing circuit during a single hyperbaric exposure. The exposure will be conducted at a partial pressure of 1.75 ATA for 240 minutes. The intervention aims to evaluate the protective effect of hydrogen gas against pulmonary oxygen toxicity.

SUMMARY:
The goal of this trial is to investigate whether adding a small fraction of hydrogen gas to an oxygen-enriched breathing mixture can reduce pulmonary oxygen toxicity (POT) in healthy and active divers from the Swedish Armed Forces. The main questions it aims to answer are:

* Does hydrogen gas reduce oxidative stress and changes in pulmonary function associated with prolonged hyperbaric oxygen exposure?
* What are the underlying pathophysiological mechanisms of pulmonary oxygen toxicity?

Researchers will compare oxygen-enriched breathing gas with 1-2% hydrogen to oxygen-enriched gas with 1-2% nitrogen (control) to see if hydrogen provides protective effects against POT during hyperbaric exposure.

Participants will:

* Complete two hyperbaric exposure sessions (hydrogen vs. nitrogen), each lasting 240 minutes at 1.75 ATA
* Undergo pulmonary function tests and sampling of blod and urin before and after each session
* Serve as their own controls in a double-blind, randomized, crossover study design

ELIGIBILITY:
Inclusion Criteria:

* Military divers actively serving, aged 20-64 years
* Meeting the Swedish Armed Forces physical standards for diving

Exclusion Criteria:

* Ongoing infection or illness that may impact pulmonary function
* Use of alcohol or smoking cigarettes within 48 hours
* Diving with any breathing gas within 48 hours
* Diving with oxygen-enriched gas (100% O₂) within 2 weeks
* Use of medications that could affect oxidative stress, lung function, or neurological status
* Medical history of serious diving-related injuries or long-term complications

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in Vital Capacity (ΔVC) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  Absolute change in vital capacity (VC), calculated as the difference in liters (L) between pre-exposure and post-exposure spirometry values, measured after each hyperbaric oxygen exposure session.

SECONDARY OUTCOMES:
Forced Expiratory Volume in One Second (FEV₁) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure
  As part of the spirometric and plethysmographic measurements, Forced Expiratory Volume in 1 second (FEV₁) will be analyzed. This represents the change (ΔFEV₁) in liters (L) between pre- and post-exposure spirometry, indicating expiratory flow capacity. Measurements follow ATS/ERS 2019 standards.
Change in FEV₁/FVC ratio | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure
  As part of the spirometric and plethysmographic measurements, the ratio between Forced Expiratory Volume in 1 second and Forced Vital Capacity (FEV₁/FVC) will be calculated. The change (ΔFEV₁/FVC) is expressed as a percentage (%) to assess airflow limitation or restriction following hyperbaric oxygen exposure.
Change in Forced Expiratory Flow 25-75% (FEF25-75%) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  As part of the spirometric and plethysmographic measurements, the mid-expiratory flow (FEF25-75%) will be assessed. This parameter reflects the mean expiratory flow between 25% and 75% of FVC and serves as an indicator of small airway function. Values are expressed in liters per second (L/s).
Change in Peak Expiratory Flow (PEF) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  As part of the spirometric and plethysmographic measurements, Peak Expiratory Flow (PEF) will be analyzed. The change (ΔPEF) represents the maximum flow achieved during forced exhalation, measured in liters per second (L/s). This outcome evaluates large airway performance.
Change in Inspiratory Capacity (IC) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  As part of the spirometric and plethysmographic measurements, Inspiratory Capacity (IC) will be determined. The change (ΔIC) in liters (L) reflects the maximal volume of air that can be inspired after a normal exhalation, providing insight into potential restrictive changes following exposure.
Change in Total Lung Capacity (TLC) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  As part of the spirometric and plethysmographic measurements, Total Lung Capacity (TLC) will be assessed. The change (Δ TLC) in liters (L) represents the total volume of air contained in the lungs after maximal inspiration, used to detect restrictive or hyperinflation patterns following hyperbaric oxygen exposure.
Residual Volume (Δ RV) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  As part of the spirometric and plethysmographic measurements, Residual Volume (RV) will be assessed. The change (Δ RV) in liters (L) represents the volume of air remaining in the lungs after maximal exhalation, used to detect gas-trapping or hyperinflation patterns associated with pulmonary oxygen toxicity
Functional Residual Capacity (Δ FRC) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  As part of the spirometric and plethysmographic measurements, Functional Residual Capacity (FRC) will be assessed. The change (Δ FRC) in liters (L) represents the volume of air remaining in the lungs at the end of a normal tidal exhalation, used to detect early alterations in lung compliance or airway closure during hyperbaric oxygen exposure.
Change in Diffusing Capacity for Carbon Monoxide (ΔDLCO) | Pre-exposure, 30-120 minutes post-exposure and 24-36 hours post-exposure.
  Absolute change in lung diffusing capacity for carbon monoxide (DLCO) , measured (mmol/min/lkPa) with single-breath DLCO test before and after each exposure, to evaluate alveolar-capillary gas exchange efficiency. DLCO values are adjusted for hemoglobin levels to improve measurement accuracy.
Airway Resistance (Impulse Oscillometry, Tremoflo™) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  Assessment of central and peripheral airway resistance (R5, R20, X5) using impulse oscillometry (Tremoflo™) before and after exposure. Evaluates small airway mechanics related to hyperbaric oxygen exposure with or without hydrogen supplementation. Unit of Measurement: cmH₂O·s/L
Index of Oxygen Stress (ΔiOS) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  Composite index derived from impulse oscillometry (Tremoflo™) representing the mean relative change from baseline in airway impedance parameters (R5, R20, X5). The Index of Oxygen Stress (iOS) quantifies oxidative stress-related changes in small airway mechanics following hyperbaric oxygen exposure with or without hydrogen supplementation.
Change in Fractional Exhaled Nitric Oxide (ΔFeNO) | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  Measurement of airway inflammation and oxidative stress via fractional exhaled nitric oxide (FeNO) levels measured in parts per billion (ppb).
Change in Exhaled Breath Particle Analysis (ΔPExA) | Pre-exposure and follow-up 24-36 hours post-exposure after each intervention.
  Change in exhaled particle count and biochemical composition (lipids, proteins, coagulation factors) reflecting epithelial lining fluid alterations.
Blood and Urinary Biomarkers of Oxidative Stress and Inflammation | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  Analysis of venous blood and urine samples for biomarkers of oxidative stress (e.g., 8-isoprostane, MDA, 8-OHdG) and inflammation (e.g., IL-6, TNF-α) to evaluate systemic effects of hyperbaric oxygen exposure with or without hydrogen supplementation. Concentrations will be quantified in standard laboratory units, for example ng/mL, pg/mL, or other equivalent measures.
Biomarkers of Neuronal Injury | Pre-exposure, 30-120 minutes post-exposure, and 24-36 hours post-exposure.
  Analysis of venous plasma samples for fluid biomarkers of neuronal injury (e.g., NfL, GFAP, Tau, UCH-L1) using NULISA™ or Simoa® HD-1 assay technologies, to evaluate central nervous system effects of hyperbaric oxygen exposure with or without hydrogen supplementation. Concentrations will be quantified in pg/mL.

OTHER OUTCOMES:
Anthropometric Measurements (Weight, Height, Sex, Age, BMI) | Baseline (Pre-exposure, prior to first dive session)
  Anthropometric data will be recorded to assess body composition and physical characteristics of the study population and to enable adjustment for potential confounders in pulmonary function outcomes. This includes body weight (kg), height (cm), biological sex (M/F), age (years), and body mass index (BMI). These variables will not serve as primary endpoints but will describe baseline characteristics and support interpretation of within-subject changes in lung function.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Blekinge Institute of Technology, Karlskrona, Blekinge County
  - Swedish Armed Forces Diving and Naval Medicine Centre (DNC), Karlskrona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] New Jersey hospital keeps detailed tracking records. OR Manager. 1989 Apr;5(4):8-9. No abstract available. PMID 10292678
- [Result] Samuels BL, Vogelzang NJ, Ruane M, Simon MA. Continuous venous infusion of doxorubicin in advanced sarcomas. Cancer Treat Rep. 1987 Oct;71(10):971-2. PMID 3652058
- [Result] Lynam C, Jennings K, Nolan K, Kane P, McKervey MA, Diamond D. Tuning and enhancing enantioselective quenching of calixarene hosts by chiral guest amines. Anal Chem. 2002 Jan 1;74(1):59-66. doi: 10.1021/ac010153k. PMID 11795818
- [Result] Ohsawa I, Ishikawa M, Takahashi K, Watanabe M, Nishimaki K, Yamagata K, Katsura K, Katayama Y, Asoh S, Ohta S. Hydrogen acts as a therapeutic antioxidant by selectively reducing cytotoxic oxygen radicals. Nat Med. 2007 Jun;13(6):688-94. doi: 10.1038/nm1577. Epub 2007 May 7. PMID 17486089

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol 2025-09-29 (2025-09-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT07263399/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocol (Updated) 2025-10-27 (2025-10-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT07263399/Prot_SAP_001.pdf